CLINICAL TRIAL: NCT02035306
Title: Usefulness of Non-invasive Pulse Co-oximetry Haemaglobin Measurements in Critically Ill Black Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chris Hani Baragwanath Academic Hospital (Other)
Collaborators: Masimo Corporation (Industry)
Responsible Party: Principal Investigator, Susan Murphy, Paediatric Intensivist, Chris Hani Baragwanath Academic Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: M120677
Record Dates: First submitted 2013-12-04; First posted 2014-01-14 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Critically Ill Black Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- non-invasive Haemaglobin (Experimental): Measuring haemaglobin using non-invasive co-oximetry device
  Interventions: Other: non invasive co-oximetry haemaglobin measurement

INTERVENTIONS:
Other: non invasive co-oximetry haemaglobin measurement

SUMMARY:
To answer the question whether a non-invasive haemaglobin measurement is clinically useful, reliable and accurate as compared to taking a blood sample and checking the haemaglobin level at the laboratory or in a blood gas analyser. This study will take place in a multi-disciplinary ICU of critically ill patients.

DETAILED DESCRIPTION:
A presenting sample of 150 patients requiring admission to ICU will be enrolled. These will include paediatric, trauma, adult medical and adult surgical patients. Informed consent will be obtained. Baseline demographic data, vital signs, Massey pigmentation score, and severity of illness scores will be calculated, as well as finger deformity, if present, nail polish or acrylics, smoking habits, finger diameter of finger measured, comorbidities and medications. Patients will be admitted in the usual way, and admission bloods will be sent to the laboratory as per usual protocol. Enrolled patients will in addition have their Haemaglobin and Plethysmography Index (measure of perfusion) measured non-invasively using the Masimo Pronto-7 handheld device. Note of concurrent medications, blood products and vital signs will be recorded at each measurement. Each patient will have measurements done 8 hourly (between 1-5 measurements per patient). Concurrent arterial blood gas samples will be taken in a heparinised syringe and performed on ABL radiometer blood gas analyser.. An additional EDTA blood sample shall be taken at each Pronto measuring point which will be measured at the laboratory on a Sysmex cell counter. Analysis of data will assess precision and accuracy, trend accuracy, and effect of pigmentation, vasopressors and other medication on the results of the non-invasive co-oximetry estimation of haemaglobin.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a condition that requires admission to ICU shall be considered to be eligible.
* Age 1month to 100years old

Exclusion Criteria:

* Patients under 1 month old
* Patients with an unrecordable blood pressure or body temperature <34 degrees.

Ages: 1 Month to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2014-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Accuracy and precision of non invasive haemaglobin measurement. | during ICU admission
  Accuracy and precision of non invasive hemoglobin (Hb) measurement to invasive co-oximetry (blood gas analyser), and laboratory haemaglobin measurement.
  For comparative purposes in our population (dark skinned patients, low Hb levels and during active transfusion) our outcome aim for Hb accuracy will be based on what Masimo has found previously in 11 335 comparisons. These are:
  * 0.99g/dl at 1SD
  * Hb between 6g/dl and 12g/dl : 95% of readings within 2g/dl of laboratory value
  * Hb between 12g/dl and 18g/dl : 95% of readings within 2g/dl of laboratory value
  Precision shall be described as a co-efficient of variation

SECONDARY OUTCOMES:
Time to result | during ICU admission
  Time to result of non invasive hemoglobin (Hb) measurement compared to invasive co-oximetry (blood gas analyser), and laboratory haemaglobin measurement (Sysmex cell counter)
Cost of test | during ICU admission
  To compare the non invasive hemoglobin (Hb) measurement to invasive co-oximetry (blood gas analyser), and laboratory haemaglobin measurement (Sysmex cell counter) with regards to cost.
Effect of skin pigmentation on result | during ICU admission
  Effect of skin pigmentation on result of non invasive hemoglobin (Hb) measurement compared to to invasive co-oximetry (blood gas analyser), and laboratory haemaglobin measurement (Sysmex cell counter)
Effect of patients clinical state on test results. | during ICU admission
  Effect of patients clinical state on test results of non invasive hemoglobin (Hb) measurement compared to invasive co-oximetry (blood gas analyser), and laboratory haemaglobin measurement (Sysmex cell counter).
  The effect of patients clinical state (temp, MAP, pH, Hb level, plethysmography index (PI), severity of illness score, presence of active transfusion, presence of active bleeding, use of pressors, use of other blood products) on test results (accuracy and precision) shall be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Chris Hani Baragwanath Hospital, Soweto, Gauteng, South Africa

REFERENCES:
- [Derived] Murphy SM, Omar S. The Clinical Utility of Noninvasive Pulse Co-oximetry Hemoglobin Measurements in Dark-Skinned Critically Ill Patients. Anesth Analg. 2018 May;126(5):1519-1526. doi: 10.1213/ANE.0000000000002721. PMID 29239951